CLINICAL TRIAL: NCT06718127
Title: Description of the Immune Response to Yellow Fever Vaccination
Acronym: IVORY2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-149
Record Dates: First submitted 2024-11-29; First posted 2024-12-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Immunization; Infections
Keywords: immunology; Vaccine response
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with an indication for primary immunization against yellow fever and typhoid (Other): People with an indication for primary immunization against yellow fever and typhoid and whose vaccination schedule includes two appointments 7 days apart
  Interventions: Biological: blood samples collection

INTERVENTIONS:
Biological: blood samples collection — blood samples collected at D0 ,W1, W5, M3 and M6

SUMMARY:
Vaccine protection depends on a specific adaptive immune memory. However, a little-explored aspect of certain live vaccines may provide beneficial, non-specific protection against infections or pathogens other than the one from which the vaccine is derived. This is the concept of innate immune memory or " trained immunity", which differs from adaptive memory in its non-specificity. Innate immune memory is triggered by exposure to immunostimulants, and offers protection against unrelated pathogenic threats for several months or even years.

The project aims to carry out an exploratory study to observe, in the context of current practice, the immune response obtained after a subunit and a live attenuated vaccine

DETAILED DESCRIPTION:
Vaccine protection depends on a specific adaptive immune memory. However, a little-explored aspect of certain live vaccines may provide beneficial, non-specific protection against infections or pathogens other than the one from which the vaccine is derived. This is the concept of innate immune memory or " trained immunity", which differs from adaptive memory in its non-specificity. Innate immune memory is triggered by exposure to immunostimulants, and offers protection against unrelated pathogenic threats for several months or even years.

For example, research has shown that the live attenuated BCG vaccine induce non-specific trained immunity, enabling innate immune cells to remember their first encounter and improve their immune status during a second confrontation with similar or different agents.

Other currently available live vaccines, such as BCG , could also "train" innate immune cells.

The project aims to carry out an exploratory study to observe, in the context of current practice, the immune response obtained after a subunit and a live attenuated vaccine

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Referred for immunisation against yellow fever and typhoid
* Any person with indication for the following vaccinations :
* Yellow fever
* Typhoïd
* Whose vaccination schedule includes two appointments 7 days apart
* Whose state of health is compatible with a single 51 ml blood sample collection
* Have consented to participate in the Ivory2 study
* Benefiting from a Social Security plan or equivalent

Exclusion Criteria:

* Anyone with a contraindication to yellow fever and/or typhoid vaccination.
* Any person who has been vaccinated against yellow fever and/or typhoid.
* Anyone who has lived in an endemic area (≥ 1 year) and/or has a history of Typhoid.
* Anyone who is unable to attend the visit 1-month after the typhoid vaccine injection.
* Women claiming to be pregnant or breast-feeding
* Anyone unable to give informed consent for participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Immunological profile of PBMCs, before and after yellow fever vaccination | 6 months
  Cytokine production assays (e.g. TNFa, IL6, IL1b)

SECONDARY OUTCOMES:
Description of the response to TyphimVi® vaccine | 6 months
  ELISA-based quantification of Anti-Vi antibody level >30 U/mL at week 5, and/or fold increase ≥2 compared with pre-vaccination IgG titer.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Taieb, Dr, Principal Investigator — Institut Pasteur
Locations (1):
- Centre Médical de l'Institut Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No